CLINICAL TRIAL: NCT02673541
Title: Randomized, Multi-Center, Comparative and Cost Effectiveness Study of a Lumen- Apposing, Covered, Self-Expanding Metal Stent (Axios™) Versus Multiple Double Pigtail Stents in the Management of Walled Off Pancreatic Necrosis
Brief Title: Study of a Lumen- Apposing, Covered, Self-Expanding Metal Stent (Axios™) Versus Multiple Double Pigtail Stents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Gardner, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D16030
Record Dates: First submitted 2016-01-11; First posted 2016-02-04 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AXIOS™ stent (Active Comparator): 1. Arm 1 will undergo EUS-guided cystogastrostomy/enterostomy and placement of the AXIOS™ stent 10-15mm (saddled diameter; choice at the discretion of the treating gastroenterologist) though the tract into the collection cavity, and correct positioning of the inner flange confirmed by EUS prior to deploying within the stomach or duodenum. Necrosectomy will be performed at the discretion of the attending gastroenterologist. Repeat endoscopy will be performed for stent removal at or before 60 days at the discretion of the attending gastroenterologist
  Interventions: Device: AXIOS™ stent
- double pigtail stents (Active Comparator): 2. Arm 2 will undergo EUS-guided cystogastrostomy/enterostomy and placement of multiple double pigtail stents (i.e. ≥2) through the tract into the collection cavity. Necrosectomy will be performed at the discretion of the attending gastroenterologist. Routine repeat treating gastroenterologist for stent removal will not be necessary, but left to the discretion of the attending gastroenterologist.
  Interventions: Device: Double Pigtail Stents

INTERVENTIONS:
Device: AXIOS™ stent — Arm 1 will undergo EUS-guided cystogastrostomy/enterostomy and placement of the AXIOS™ stent 10-15mm (saddled diameter; choice at the discretion of the treating gastroenterologist) though the tract into the collection cavity, and correct positioning of the inner flange confirmed by EUS prior to deploying within the stomach or duodenum.
  Arms: AXIOS™ stent
Device: Double Pigtail Stents — Arm 2 will undergo EUS-guided cystogastrostomy/enterostomy and placement of multiple double pigtail stents (i.e. ≥2) through the tract into the collection cavity.
  Arms: double pigtail stents

SUMMARY:
The present study aims to compare the clinical efficacy and cost effectiveness of the AXIOS™ stent versus the "conventional" approach using double pigtail plastic stents in the treatment of patients with walled-off pancreatic necrosis.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is responsible for nearly a quarter million hospital admissions annually and will affect around 40 per 100,000 persons per year (1). The majority of patients experience a clinically mild course; however, as many as one in five patients develop a severe illness associated with a high mortality (2). In early phases of the disease, there is an acute inflammatory process that may involve necrosis of the pancreatic or peri-pancreatic tissues (3). There are also delayed complications that may develop locally, usually over a period of weeks, which include the formation of walled-off fluid collections. These are sometimes composed of simple fluid and termed pseudocysts, while in other cases they represent organization and encapsulation of sterile or infected necrosis and are termed walled-off pancreatic necrosis (WOPN) (4). The indication to drain or debride these collections usually depends upon on a number of factors, but principally on whether they are symptomatic, infected, or responsible for other local or systemic complications.

The contemporary management strategy for walled-off pancreatic fluid collections has shifted in recent years. Surgery, and even percutaneous catheter drainage, should no longer be considered the initial mainstay of therapy in place of endoscopic drainage for simple pseudocysts (5) (6). In addition there is good evidence to support an endoscopic approach for patients with infected necrosis (7). There are now numerous publications reporting the success of direct endoscopic transmural drainage or necrosectomy (ETD/N) for a variety of indications including infected and sterile walled-off collections (8).

The issue that now deserves attention is a matter of selecting the best technique to accomplish ETD/N. The current process involves first creating a cystenterostomy to gain access to the walled-off collection, dilating the tract, and then inserting a drainage device. However, there are a variety of available devices and methods in use for drainage, and to our knowledge, none to date have been directly compared in a randomized controlled trial.

The conventional approach involves inserting either a pair or more of plastic double pigtail stents or a self-expanding metal stent (SEMS) through a cystenterostomy: both approaches have limitations, and may require multiple endoscopic sessions before definitive resolution (9). One, the pigtail stents have a narrow lumen (7F-10F) and often migrate or become occluded (10). Two, the SEMS also have a tendency occlude, cause local trauma with bleeding and infection, and migrate, which has led some to also use double pigtails to help anchor the SEMS in place (11) (12).

These challenges have led to the innovation of large caliber covered stents with flanges on either end to facilitate apposition of the cyst wall and enteral tissues, preventing migration, and allowing for necrosectomy through their wide lumen. To our knowledge there are at least two designs in production; the AXIOS™ stent and the Nagi stent (13) (14). There is now a fair amount of experience, particularly using the AXIOS™ stent (with or without a novel NAVIX access system) for both WOPN and pseudocysts, with the majority of reports showing it to be safe and effective (15) (16) (17) (18) (19) (20). The device has also been successfully used for novel indications including access and drainage of the gallbladder and an intrathoracic fluid collection (21) (22) (23). The AXIOS™ stent is FDA approved for the indication of draining walled off pancreatic necrosis.

The present study aims to compare the clinical efficacy and cost effectiveness of the AXIOS™ stent versus the "conventional" approach using double pigtail plastic stents in the treatment of patients with walled-off pancreatic necrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18-80 years old (including patients aged 18 and 80)
2. Subjects capable of giving informed consent
3. Patients carrying the diagnosis or symptomatic sterile or infected walled-off pancreatic necrosis (WOPN) based upon Atlanta Classification (4) ≥ 4cm in largest diameter, deemed to require and amenable to endoscopic transmural drainage with or without necrosectomy by attending gastroenterologist
4. Fluid collection size ≥ 4cm in largest diameter (based on CT, MRI, transabdominal or endoscopic ultrasound within 30days)
5. Fluid collection that is adherent to the stomach/bowel wall allowing for fistula tract creation
6. Fluid collection containing significant amount of necrotic material (defined as >30% of echogenic material by ultrasound/EUS, or necrotic debris by CT/MRI)

Exclusion Criteria:

1. Inability to provide written informed consent
2. Contraindications to endoscopic treatment as determined by the gastroenterologist attending
3. Pregnant or nursing mothers
4. Bleeding or coagulation disorder
5. Previous surgical or endoscopic cystogastrostomy/enterostomy or necrosectomy
6. Shock
7. Cystic neoplasms or pancreatic malignancy
8. Pseudocysts
9. Subjects cannot be homeless or incarcerated
10. Age younger than 18 or older than 80
11. More than one pancreatic/peri-pancreatic fluid collection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gardner, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Whitcomb DC. Clinical practice. Acute pancreatitis. N Engl J Med. 2006 May 18;354(20):2142-50. doi: 10.1056/NEJMcp054958. No abstract available. PMID 16707751
- [Background] Acevedo-Piedra NG, Moya-Hoyo N, Rey-Riveiro M, Gil S, Sempere L, Martinez J, Lluis F, Sanchez-Paya J, de-Madaria E. Validation of the determinant-based classification and revision of the Atlanta classification systems for acute pancreatitis. Clin Gastroenterol Hepatol. 2014 Feb;12(2):311-6. doi: 10.1016/j.cgh.2013.07.042. Epub 2013 Aug 16. PMID 23958561
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Varadarajulu S, Bang JY, Sutton BS, Trevino JM, Christein JD, Wilcox CM. Equal efficacy of endoscopic and surgical cystogastrostomy for pancreatic pseudocyst drainage in a randomized trial. Gastroenterology. 2013 Sep;145(3):583-90.e1. doi: 10.1053/j.gastro.2013.05.046. Epub 2013 May 31. PMID 23732774
- [Background] Johnson MD, Walsh RM, Henderson JM, Brown N, Ponsky J, Dumot J, Zuccaro G, Vargo J. Surgical versus nonsurgical management of pancreatic pseudocysts. J Clin Gastroenterol. 2009 Jul;43(6):586-90. doi: 10.1097/MCG.0b013e31817440be. PMID 19077728
- [Background] Bakker OJ, van Santvoort HC, van Brunschot S, Geskus RB, Besselink MG, Bollen TL, van Eijck CH, Fockens P, Hazebroek EJ, Nijmeijer RM, Poley JW, van Ramshorst B, Vleggaar FP, Boermeester MA, Gooszen HG, Weusten BL, Timmer R; Dutch Pancreatitis Study Group. Endoscopic transgastric vs surgical necrosectomy for infected necrotizing pancreatitis: a randomized trial. JAMA. 2012 Mar 14;307(10):1053-61. doi: 10.1001/jama.2012.276. PMID 22416101
- [Background] Haghshenasskashani A, Laurence JM, Kwan V, Johnston E, Hollands MJ, Richardson AJ, Pleass HC, Lam VW. Endoscopic necrosectomy of pancreatic necrosis: a systematic review. Surg Endosc. 2011 Dec;25(12):3724-30. doi: 10.1007/s00464-011-1795-x. Epub 2011 Jun 9. PMID 21656324
- [Background] Talreja JP, Shami VM, Ku J, Morris TD, Ellen K, Kahaleh M. Transenteric drainage of pancreatic-fluid collections with fully covered self-expanding metallic stents (with video). Gastrointest Endosc. 2008 Dec;68(6):1199-203. doi: 10.1016/j.gie.2008.06.015. PMID 19028232
- [Background] Wrobel PS, Kaplan J, Siddiqui AA. A new lumen-apposing metal stent for endoscopic transluminal drainage of peripancreatic fluid collections. Endosc Ultrasound. 2014 Oct;3(4):203-4. doi: 10.4103/2303-9027.144508. No abstract available. PMID 25485266
- [Background] Paradigm shift away from open surgical necrosectomy toward endoscopic interventions for necrotizing pancreatitis. Jae Hee Cho, Yoon Jae Kim, and Yeon Suk Kim. s.l. : Gastrointestinal Intervention 2014; 3(2): 84-88.
- [Background] Chaves DM, Monkemuller K, Carneiro F, Medrado B, Dos Santos M, Wodak S, Reimao S, Sakai P, de Moura E. Endoscopic treatment of large pancreatic fluid collections (PFC) using self-expanding metallic stents (SEMS) - a two-center experience. Endosc Int Open. 2014 Dec;2(4):E224-9. doi: 10.1055/s-0034-1390796. Epub 2014 Oct 29. PMID 26135097
- [Background] Yamamoto N, Isayama H, Kawakami H, Sasahira N, Hamada T, Ito Y, Takahara N, Uchino R, Miyabayashi K, Mizuno S, Kogure H, Sasaki T, Nakai Y, Kuwatani M, Hirano K, Tada M, Koike K. Preliminary report on a new, fully covered, metal stent designed for the treatment of pancreatic fluid collections. Gastrointest Endosc. 2013 May;77(5):809-14. doi: 10.1016/j.gie.2013.01.009. Epub 2013 Feb 26. PMID 23453183
- [Background] Shah RJ, Shah JN, Waxman I, Kowalski TE, Sanchez-Yague A, Nieto J, Brauer BC, Gaidhane M, Kahaleh M. Safety and efficacy of endoscopic ultrasound-guided drainage of pancreatic fluid collections with lumen-apposing covered self-expanding metal stents. Clin Gastroenterol Hepatol. 2015 Apr;13(4):747-52. doi: 10.1016/j.cgh.2014.09.047. Epub 2014 Oct 5. PMID 25290534
- [Background] Gornals JB, De la Serna-Higuera C, Sanchez-Yague A, Loras C, Sanchez-Cantos AM, Perez-Miranda M. Endosonography-guided drainage of pancreatic fluid collections with a novel lumen-apposing stent. Surg Endosc. 2013 Apr;27(4):1428-34. doi: 10.1007/s00464-012-2591-y. Epub 2012 Dec 12. PMID 23232994
- [Background] Binmoeller KF, Smith I, Gaidhane M, Kahaleh M. A kit for eus-guided access and drainage of pancreatic pseudocysts: efficacy in a porcine model. Endosc Ultrasound. 2012 Oct;1(3):137-42. doi: 10.7178/eus.03.004. PMID 24949351
- [Background] 141 EUS-Guided Drainage of Pancreatic Pseudocysts (PP) Utilizing a Novel Anchoring, Covered Self-Expanding Metal Stent (Acsems): Results From a Prospective, Multi-Center Study. Shah, Raj J. et al. s.l. : Gastrointestinal Endoscopy , Volume 77 , Issue 5 , AB128 .
- [Background] Gornals JB, Parra C, Pelaez N, Secanella L, Ornaque I. Double endosonography-guided transgastric and transduodenal drainage of infected pancreatic-fluid collections using metallic stents. Rev Esp Enferm Dig. 2013 Mar;105(3):163-5. doi: 10.4321/s1130-01082013000300007. No abstract available. PMID 23735023
- [Background] Binmoeller KF, Shah J. A novel lumen-apposing stent for transluminal drainage of nonadherent extraintestinal fluid collections. Endoscopy. 2011 Apr;43(4):337-42. doi: 10.1055/s-0030-1256127. Epub 2011 Jan 24. PMID 21264800
- [Background] Itoi T, Binmoeller KF, Shah J, Sofuni A, Itokawa F, Kurihara T, Tsuchiya T, Ishii K, Tsuji S, Ikeuchi N, Moriyasu F. Clinical evaluation of a novel lumen-apposing metal stent for endosonography-guided pancreatic pseudocyst and gallbladder drainage (with videos). Gastrointest Endosc. 2012 Apr;75(4):870-6. doi: 10.1016/j.gie.2011.10.020. Epub 2012 Jan 31. PMID 22301347

RESULTS

PARTICIPANT FLOW:
Groups:
- AXIOS™ Stent: Arm 1 will undergo EUS-guided cystogastrostomy/enterostomy and placement of the AXIOS™ stent 10-15mm (saddled diameter; choice at the discretion of the treating gastroenterologist) through the tract into the collection cavity, and correct positioning of the inner flange confirmed by EUS prior to deploying within the stomach or duodenum. Necrosectomy will be performed at the discretion of the attending gastroenterologist. Repeat endoscopy will be performed for stent removal at or before 60 days at the discretion of the attending gastroenterologist
- Double Pigtail Stents: Arm 2 will undergo EUS-guided cystogastrostomy/enterostomy and placement of multiple double pigtail stents (i.e. ≥2) through the tract into the collection cavity. Necrosectomy will be performed at the discretion of the attending gastroenterologist. Routine repeat treating gastroenterologist for stent removal will not be necessary, but left to the discretion of the attending gastroenterologist.
  Double Pigtail Stents: Arm 2 will undergo EUS-guided cystogastrostomy/enterostomy and placement of multiple double pigtail stents (i.e. ≥2) through the tract into the collection cavity.
Period: Overall Study
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AXIOS™ Stent: Arm 1 will undergo EUS-guided cystogastrostomy/enterostomy and placement of the AXIOS™ stent 10-15mm (saddled diameter; choice at the discretion of the treating gastroenterologist) though the tract into the collection cavity, and correct positioning of the inner flange confirmed by EUS prior to deploying within the stomach or duodenum. Necrosectomy will be performed at the discretion of the attending gastroenterologist. Repeat endoscopy will be performed for stent removal at or before 60 days at the discretion of the attending gastroenterologist
- Total: Total of all reporting groups
Arm/Group | AXIOS™ Stent | Double Pigtail Stents | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 46 (2) | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Cost Differences
Description: To compare the cost differences of the AXIOS™ stent vs. multiple double pigtail stents in the management of walled-off pancreatic necrosis.
Time Frame: Subject followed for an average of one year
Population: data was not collected or analyzed
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Definitive Resolution
Description: 1. To compare the relative efficacy in terms of definitive resolution of walled off pancreatic necrosis using the AXIOS™ stent vs. multiple double pigtail stents.
Time Frame: Subject followed for an average of one year
Measure: Number; unit: participants
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
Number analyzed (Participants) | 3 | 2
participants | 1 | 1
Statistical Analysis 1: Comparison: AXIOS™ Stent vs Double Pigtail Stents; Test type: Other; p = 1, Fisher Exact

3. Secondary Outcome: Number of Endoscopic Sessions
Description: 2. To compare the number of endoscopic sessions required to achieve definitive resolution of walled-off pancreatic fluid necrosis using the AXIOS™ stent vs. multiple double pigtail stents.
Time Frame: Subject followed for an average of one year
Population: Data not collected
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Additional Procedures
Description: 3. To compare the number of additional procedures (surgical, percutaneous, or nasocystic) required to achieve definitive resolution of walled-off pancreatic necrosis using the AXIOS™ stent vs. multiple double pigtail stents.
Time Frame: Subject followed for an average of one year
Population: data not collected
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Frequency of Stent Migration
Description: 4. To compare the frequency of stent migration using the AXIOS™ stent vs. multiple double pigtail stents in the management of walled-off pancreatic necrosis.
Time Frame: Subject followed for an average of one year
Population: data not collected
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events
Description: 5. To compare the safety and tolerability of the AXIOS™ stent vs. multiple double pigtail stents in the management of walled-off pancreatic necrosis as assessed by the collected of adverse events over the course of the study, including but not limited to: bleeding, infections, stent migration, surgery and pain.
Time Frame: Subject followed for an average of one year
Population: details of the adverse events are in the adverse events section
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
Number analyzed (Participants) | 3 | 2
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | AXIOS™ Stent | Double Pigtail Stents
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS™ Stent (N=3) | Double Pigtail Stents (N=2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS™ Stent (N=3) | Double Pigtail Stents (N=2)
MIld/moderate bleeding (Gastrointestinal disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT02673541/Prot_SAP_000.pdf